CLINICAL TRIAL: NCT01775007
Title: A Pilot Study to Test the Safety and Feasibility of a Brillouin Ocular Analyzer
Acronym: Brillouin I
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Seok Hyun Yun, Associate Physicist / Associate Professor, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 2008-P-002176/10
Record Dates: First submitted 2013-01-22; First posted 2013-01-24 (Estimated); Last update posted 2022-08-02 (Actual); Status verified 2022-07

CONDITIONS: Measurement of the Elasticity of the Anterior Eye Segment
Keywords: Lens; Cornea; Presbyopia
MeSH Terms: conditions — Corneal Diseases; Presbyopia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Normal Healthy Subjects (Experimental): Brillouin Ocular Analyser
  Interventions: Device: Brillouin Ocular Analyser

INTERVENTIONS:
Device: Brillouin Ocular Analyser — Measurement of the local viscoelastic properties (Brillouin Shift) of the Anterior Eye Segment.

SUMMARY:
A Brillouin ocular analyzer uses a low-power near infrared laser light to probe the viscoelastic properties of the cornea and crystalline lens in the eye. The study hypothesis is that the instrument can measure the Brillouin light scattering spectra from the eye safely and effectively from human subjects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers aged 20-60
* No refractional abnormalities
* Clear enough cornea and media to permit imaging

Exclusion Criteria:

* Occludable narrow angles (without a patent peripheral iridotomy)
* Other ocular or systemic pathology, which precludes safe eye dilation
* LASIK eye surgery
* Allergies to the dilation medication
* Only one healthy eye
* Pregnant women or expected pregnancy within the timeframe of the study
* Do not or cannot understand the instructions for the imaging
* Restricted mobility

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 31 (Actual)
Dates: Start 2011-03 (Actual); Primary Completion 2017-09 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
Number of patients with adverse events | 6 months
  Complete standard eye exam including medical and ocular history with manifest refraction, Amsler grid evaluation (macular test), color vision (Ishihara color plates), Scotopic pupil measurement (Colvard pupillometer), Slit lamp biomicroscopy of anterior segment, intraocular pressure measurement, dilated fundoscopic exam (2.5% phenylephrine and 0.5% tropicamide), and corneal topography (Pentacam).

SECONDARY OUTCOMES:
Sensitivity and accuracy of Brillouin modulus measurement. | at time of imaging session
  It will be tested if, with the parameters designed for in vivo operation, the Brillouin ocular analyzer is sensitive enough to characterize the elasticity of cornea and crystalline lens as well as its spatial distribution within the ocular tissue.

CONTACTS AND LOCATIONS:
Overall Officials: Seok-Hyun Yun, PhD, Principal Investigator — Massachusetts General Hospital
Locations (2):
- United States (2):
  - Massachusetts Eye and Ear Infirmary, Boston, Massachusetts
  - Massachusetts General Hospital, Boston, Massachusetts

REFERENCES:
- [Result] Scarcelli G, Yun SH. In vivo Brillouin optical microscopy of the human eye. Opt Express. 2012 Apr 9;20(8):9197-202. doi: 10.1364/OE.20.009197. PMID 22513631